CLINICAL TRIAL: NCT05612256
Title: Electrical Impedance Tomography for Identification of Optimal Positive End-expiratory Pressure in Newborn Infants
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-00508; ks22Gerull
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Positive End-expiratory Pressure (PEEP)
Keywords: respiratory support; newborn infants; ventilator induced lung injury (VILI); mechanical ventilation; electrical impedance tomography (EIT); forced oscillation technique (FOT); saturation oxygenation pressure index (SOPI); ventilation to perfusion ratio; regional lung ventilation patterns; Silent Spaces
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants on mechanical ventilation
  Interventions: Diagnostic Test: Electrical impedance tomography (EIT); Diagnostic Test: Forced oscillation technique (FOT); Diagnostic Test: Saturation oxygenation pressure index (SOPI)
- Infants on non-invasive respiratory support
  Interventions: Diagnostic Test: Electrical impedance tomography (EIT); Diagnostic Test: Saturation oxygenation pressure index (SOPI)

INTERVENTIONS:
Diagnostic Test: Electrical impedance tomography (EIT) — EIT is the measurement of impedance changes of the lung against the flow of alternating electrical currents applied to the thorax. The signal of the electrodes is transmitted to a monitor, which enables real-time assessment of lung aeration and changes in lung volume. EIT is able to reconstruct impedance changes with a high temporal resolution and allows calculation of tidal volumes, relative stretch of lung tissue and areas of poor ventilation. Areas with impedance changes of < 10 % of the maximum impedance changes are called 'Silent Spaces'.
Diagnostic Test: Forced oscillation technique (FOT) — FOT enables non-invasive assessment of lung mechanics using sound waves to inform about the respiratory impedance of the respiratory system (Zrs). Reactance of the respiratory system (Xrs) as part of Zrs is a surrogate measure of compliance of the respiratory system. Xrs was previously used to identify optimal PEEP level, i.e., the PEEP at highest compliance equivalent, in newborn infants using a setup requiring research-specific hardware and software. The FOT module integrated in the commercially available neonatal ventilator is routinely used. FOT measurements are performed twice at each PEEP level to assess the reproducibility of the measurements.
  Groups: Infants on mechanical ventilation
Diagnostic Test: Saturation oxygenation pressure index (SOPI) — SOPI is assessed non-invasively and calculated from standard monitoring parameters such as PEEP, fraction of inspired oxygen pressure (FiO2) and peripheral oxyhaemoglobin saturation (SpO2) (PEEP x FiO2 x 100) / SpO2). SOPI is used to provide information on ventilation to perfusion ratio dependent on PEEP level.

SUMMARY:
Electrical impedance tomography (EIT) enables assessment of regional lung ventilation at the bedside. EIT has been safely used in newborn infants to image intrathoracic lung volume patterns as early as from the first minute of life. This prospective single-centre observational study is to identify optimal PEEP in infants on respiratory support by measurements of EIT, FOT and SOPI.

DETAILED DESCRIPTION:
Evidence-based guidelines on the optimal level of positive end-expiratory pressure (PEEP) in newborn infants on respiratory support do not exist. Furthermore, there is a lack of simple bed-side parameters to guide clinicians towards the optimal PEEP level. Nevertheless, PEEP requires individual adjustment to minimize ventilator induced lung injury (VILI), shorten the duration of mechanical ventilation and reduce respiratory long-term morbidity.

Potential techniques to assess optimal PEEP level in infants on respiratory support include electrical impedance tomography (EIT), the forced oscillation technique (FOT) and the saturation oxygenation pressure index (SOPI). EIT is a promising non-invasive technique that provides information on regional changes in lung aeration and ventilation inhomogeneity. FOT is used in mechanically ventilated or spontaneously breathing infants and provides information on reactance (Xrs) and resistance (Rrs) of the respiratory system. SOPI is a score calculated from the PEEP level, the amount of administered oxygen (FiO2) and the infant's peripheral oxyhaemoglobin saturation (SpO2). SOPI provides information on the ventilation to perfusion ratio dependent on the PEEP level. EIT, FOT and SOPI seem promising tools for identification of optimal PEEP in newborn infants on respiratory support. In particular, a combination of information on regional ventilation (by EIT), global lung mechanics (by FOT) and ventilation to perfusion ratio (by SOPI) will improve the understanding of optimal PEEP and may reduce long-term respiratory sequelae.

This prospective single-centre observational study is to identify optimal PEEP in infants on respiratory support by measurements of EIT, FOT and SOPI. Measurements are performed once daily during the first three days on respiratory support and are repeated in weekly intervals if the infant remains mechanically ventilated. An additional measurement is planned after extubation.

ELIGIBILITY:
Inclusion Criteria:

* 22+0 to 41+6 weeks' gestational age
* Requiring mechanical ventilation
* Written informed parental consent

Exclusion Criteria:

* Major congenital malformations including lung and cardiac malformations
* Infants on high frequency oscillatory ventilation
* Lack of written informed parental consent

Ages: 0 Days to 28 Days | Sex: All
Age Groups: Child
Study Population: All newborn infants admitted to the University Children's Hospital Basel UKBB requiring mechanical ventilation are eligible for the study.
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in composite score consisting of proportionally weighted raw values of Silent Spaces, Xrs and SOPI (mechanical ventilation) | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  A composite score consisting of proportionally weighted raw values of Silent Spaces, respiratory reactance (Xrs) and SOPI (mechanical ventilation)
Change in composite score consisting of proportionally weighted raw values of Silent Spaces and SOPI (non-invasive respiratory support) | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  A composite score consisting of proportionally weighted raw values of Silent Spaces and SOPI (non-invasive respiratory support)
Change in Silent Spaces (areas of atelectasis as well as overdistension) | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  Silent Spaces measured by EIT (calculated from electrical impedance)
Change in respiratory reactance (Xrs) (measure of compliance of the respiratory system) | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  Respiratory reactance reflects inertance and compliance of the lungs and can be viewed as rebound resistance
Change in Saturation oxygenation pressure index (SOPI) | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  Calculated from standard monitoring parameters such as PEEP, fraction of inspired oxygen pressure (FiO2) and peripheral oxyhaemoglobin saturation (SpO2) (PEEP x FiO2 x 100) / SpO2)

SECONDARY OUTCOMES:
Change in Delta impedance (ΔZ) | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  Delta impedance (ΔZ) is an additional EIT parameter
Change in centre of ventilation (CoV) | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  Centre of ventilation (CoV) is an additional EIT parameter
Change in tidal volume (VT,EIT) | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  Tidal volume (VT,EIT) is an additional EIT parameter
Change in driving pressure of the respiratory system (Peak plateau pressure - PEEP) | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
Change in resistance (Rrs) of the respiratory system | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  Resistance (Rrs) is an additional FOT parameter
Change in peak inspiratory pressure | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  Peak inspiratory pressure is a mechanical ventilation parameters
Change in tidal volume per kg body weight (VT/kg) | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  Tidal volume per kg body weight (VT/kg) is a mechanical ventilation parameters
Change in dynamic compliance | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  Dynamic compliance is a mechanical ventilation parameters
Change in respiratory rate | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)
  Respiratory rate is a mechanical ventilation parameters
Change in transcutaneous CO2 pressure (tcpCO2) | Once daily during the first three days on respiratory support and weekly intervals if the infant remains mechanically ventilated (approx. 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Gerull, Dr. med., Principal Investigator — Department of Neonatology, University Children's Hospital Basel UKBB
Locations (1):
- Department of Neonatology, University Children's Hospital Basel UKBB, Basel, Switzerland